CLINICAL TRIAL: NCT01091909
Title: Post-extraction Wound Healing in Patients With Type 2 Diabetes
Acronym: PEWHPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Karin Sa Fernandes, PhD student, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FR- 225568
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; wound healing; neutrophil count; dental extraction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tooth Extraction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- post-extraction wound healing (Experimental): 53 individuals with diabetes and 29 controls, without diabetes, were followed for 60 days after dental extractions, and were examined after 3, 7, 21, and 60 postoperative days.
  Interventions: Procedure: Dental extractions

INTERVENTIONS:
Procedure: Dental extractions — All dental extractions were performed at an outpatient clinic at the USP Dental School. In addition, all extractions were performed under local anesthesia by the same experienced dentist, in accordance with the standards established by Peterson et al (2008).

SUMMARY:
The purpose of this study is to evaluate clinical healing after dental extraction and the occurrence of surgical complications in patients with type 2 diabetes and compare with non-diabetic patients or control, taking into account laboratory data such as blood count, glycated hemoglobin (HbA1) and immunological profile of the patients.

DETAILED DESCRIPTION:
It has been established in scientific literature that patients with diabetes have a greater predisposition to oral complications and that oral infections may compromise their metabolic control. There is scant clinical evidence of a relationship between diabetes and an increased risk of infection after dental extractions. To our knowledge, no prospective longitudinal studies have been designed to prove this hypothesis.

The aim of this study is to evaluate clinical healing after dental extraction and the occurrence of surgical complications in patients with type 1 and 2 diabetes and compare with non-diabetic patients, taking into account laboratory data such as blood count, glycated hemoglobin (HbA1) and immunological profile of the patients.

Ninety patients shall be prospectively studied, divided into 3 groups: Group 1 will consist of 30 patients with uncontrolled type 2 diabetics patients, group 2 will consist of 30 controlled type 2 diabetics patients and group 3 composed of 30 non-diabetic patients (control group).

All patients will undergo extraction of erupted teeth, always carried out by the same dentist (MS).

A complete medical history and laboratory tests will be conducted for all patients including: glycated hemoglobin (HbA1), fasting glucose, complete blood count, platelets, prothrombin time (PT), partial thromboplastin time (PTT), immunoglobulins (IgA, IgG and IgM), CD3, CD4, CD8, testing of complement (C3, C4), dihydrorhodamine (DHR) oxidation, phagocytosis index test and neutrophil chemotaxis.

At the end of surgery, blood pressure and plasma glucose by finger prick will be measured again. Surgery characteristics will be recorded, such as: length of surgery time from anesthesia to sutures, whether forceps and/or lever were used, the need to use a flap approach, the number of vials of anesthetic used, and intra-ligament anesthesia.

The clinical assessment of healing will take place 3, 7, 21, and 60 days after surgery and will be performed by the same dentist who perform the surgeries (KSF), blinded to the group of the patient and laboratory exams. On these days, the region will be examined, photographed and will be applied to the Visual Analogic Scale (VAS).

On day 60 after surgery, the postoperative period will be classified as: 1) no complications or 2) with complications, according to Cheung et al 2001. The following situations will be considered as complications after dental extraction:

1. Acute infection of the alveolus: pain, erythema, edema, purulent discharge and fever;
2. Acute inflammation of the alveolus: pain, inflamed alveolar tissue, absence of pus and fever;
3. Dry socket: persistent pain and exposure of the alveolar bone.

All this clinical information will determine the post-operative quality regarding the healing time and occurrence of infection and inflammation of the alveoli.

Data will be statistically analyzed in order for us to understand the pattern of healing and occurrence of complications after dental extraction in the studied groups. The data analyzed will include hematological data, immunological profile and the glycated hemoglobin of patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be treated at the dental clinic of CAPE-FOUSP (Special Care Dentistry Center, School of Dentistry, University of São Paulo), and will be selected for the study when they require simple extraction of the first or second lower molar.

Exclusion Criteria:

* Patients that will be excluded from both groups are those who come to the clinic in an emergency dental situation, those who are using (or have used within one month previous) hormones, antibiotics, anti-inflammatory drugs, bisphosphonates, smokers, drug users and chronic alcohol users. Patients with thyroid disorders and those who are unable to measure capillary blood glucose at home will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-03; Primary Completion 2013-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 3, 7, 21, and 60 postoperative days
  Postoperative complications included the following signs and symptoms: edema; erythema; alveolar bone exposure; halitosis; trismus; fever; cellulitis; Ludwig's angina; loss of appetite; malaise; itching; moderate pain (as assessed by a visual analog scale); and unpleasant taste.

SECONDARY OUTCOMES:
Delayed wound healing | 3, 7, 21, and 60 postoperative days
  According to the literature, the dental alveolus is filled with blood clot and fibrin at 3 days after dental extraction; on postoperative day 7, the alveolus is filled with granulation tissue; on postoperative day 21, wound epithelialization is complete; and on postoperative day 60, alveolar bone formation can be observed on a dental radiographic image. Delayed wound healing was defined as a delay in any of the aforementioned events.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Gallottini, PhD, Study Chair — Head of the Special Care Dentistry Center of Dental School of University of Sao Paulo
Locations (1):
- School of Dentistry of University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Barasch A, Safford MM, Litaker MS, Gilbert GH. Risk factors for oral postoperative infection in patients with diabetes. Spec Care Dentist. 2008 Jul-Aug;28(4):159-66. doi: 10.1111/j.1754-4505.2008.00035.x. PMID 18647376
- [Background] Bergman SA. Perioperative management of the diabetic patient. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Jun;103(6):731-7. doi: 10.1016/j.tripleo.2006.11.029. Epub 2007 Mar 26. PMID 17376713